CLINICAL TRIAL: NCT05981651
Title: Development and Application of a Dynamic Three-dimensional Quantitative Facial Measurement Device
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Guodong Feng, chief physician, Peking Union Medical College Hospital
Other Study IDs: PekingUMCH record I-22PJ1121
Record Dates: First submitted 2023-07-27; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Facial Palsy
MeSH Terms: conditions — Facial Paralysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- training session: A total of 150 facial expression videos of healthy volunteers and facial palsy patients were collected as a training set for the algorithm
  Interventions: Other: non-intervention
- test set: A total of 50 cases of healthy volunteers and patients with facial palsy were used as the test set for the algorithm
  Interventions: Other: non-intervention

INTERVENTIONS:
Other: non-intervention — non-intervention

SUMMARY:
The aim of this project is to successfully develop and industrialise the "Facial Movement 3D Dynamic Quantitative Measurement Device", which is a commercial device that can provide dynamic indicators of facial movement, and can practically solve the evaluation problems of facial paralysis for doctors and patients, and has important clinical value and social benefits.

DETAILED DESCRIPTION:
Based on the current optimal high-precision face key point technology, the effective high-precision automatic face recognition model conforming to the Asian face is established through specialised training with targeted marker data, time series training optimisation based on optical flow, and local image tracking technology. The 3D reconstruction technique is then used to reconstruct the 3D spatial coordinates of the face keypoints, so as to realise the multi-camera 3D tracking of the face keypoints. The displacement of the key points is used to respond to the facial muscle activity characteristics of facial paralysis patients.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 14 years
2. No history of facial surgery, facial trauma, or scars obscuring the facial features.
3. Able to perform relevant actions according to instructions
4. Willingness to participate in the study

Exclusion Criteria:

1. Unwillingness to participate in the study
2. Unable to co-operate with relevant command actions
3. Obvious trauma, scars, etc. obscuring the facial features
4. Less than 14 years of age

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Based on previous face data collection often use larger public datasets, such as the AFLW dataset with 20,000 images. we need the same order of magnitude of local ethnographic data for migration learning. At the same time, the data in the dataset is improved according to the need to improve the accuracy of the labelled data at key points. Take about 100 effective frames for each data set. Need to complete about 200 people of various types of face data acquisition. The test group data is generally designed to be more than 20% of the training data, so the number of test group samples is designed to be 50 groups.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Facial feature point displacement distance | 3 months
  Displacement of corresponding facial feature points when volunteers perform specific actions such as specific expressions (raising eyebrow, closing eyes, shrugging nose, smiling and whistling)
Facial Feature Point Velocity | 3 months
  Velocity of the corresponding facial feature points of volunteers when accomplishing specific actions such as specific expressions (raising eyebrows, closing eyes, shrugging nose, smiling, whistling)

CONTACTS AND LOCATIONS:
Overall Officials: Guodong Feng, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No